CLINICAL TRIAL: NCT03278262
Title: INSIGHT - The Impact of baseliNe viSual Acuity on the Treatment Outcomes in Patients Treated With AflIbercept in Real-life Clinical settinG. Analysis of Data From the SwedisH Macula RegisTer
Brief Title: The Impact of Baseline Visual Acuity on the Treatment Outcomes in Patients Treated With AflIbercept in Real-life Clinical Setting
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 19473
Record Dates: First submitted 2017-08-28; First posted 2017-09-11 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- >= 70 letters: Baseline VA >= 70 letters
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- 36-69 letters: Baseline VA 36-69 letters
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- <=35 letters: Baseline VA <=35 letters
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Treatment-naïve eyes with neovascularization AMD (Age-related Macular Degeneration), with the indication to be treated with Aflibercept. One and/or two eyes per patient.

SUMMARY:
The study will assess the mean change in Visual Acuity (VA) (overall and stratified by baseline VA) at year 1 and 2 of treatment with Aflibercept in real-life setting.

In addition, the study will ascertain the baseline VA in treatment -naïve Wet Age-Related Macular Degeneration or neo-vascular AMD (wAMD) patients who start treatment with Aflibercept in a real-life setting and it will assess the impact of baseline VA on the outcomes of Aflibercept treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve eyes with neovascularization AMD, with the indication to be treated with Aflibercept. One and/or two eyes per patient.

Exclusion Criteria:

* Eyes treated previously with another anti-VEGF drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in the Swedish Macula Register during the study period.
Sampling Method: Probability Sample
Enrollment: 2312 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Visual Acuity (VA) (Snellen) | at 3±1 months, 6±1months, 12±2 months and at 24±2 months follow-up
  Change in VA (Snellen) at 3±1 months, 6±1months, 12±2 months and at 24±2 months follow-up in all eyes and stratified in the three groups by Visual Acuity (VA) at baseline.
Change in Early Treatment Diabetic Retinopathy Study (ETDRS) | at 3±1 months, 6±1months, 12±2 months and at 24±2 months follow-up
  Change Early Treatment Diabetic Retinopathy Study (ETDRS) in all eyes and stratified in the three groups by VA at baseline.
Change in Lasbarhetsindex (LIX, Readability Index) | at 3±1 months, 6±1months, 12±2 months and at 24±2 months follow-up
  Change in LIX in all eyes and stratified in the three groups by VA at baseline. LIX: Jaeger/LIX adult A chart (Ortho-KM, Lund, Sweden). The LIX-chart is a standardized readability index for measuring near vision and it is used almost ubiquitously in eye clinics in Sweden

SECONDARY OUTCOMES:
Proportion of patients with Gain of vision 5 to 15 letters; > 15 letters; Loss of vision >5 to <15 letters; >15 letters or Stable -5 to +5 letters at the annual time points | At year 1 and year 2
  Patients with Gain of vision 5-15 letters, > 15 letters; Loss of vision >5-<15 letters; >15 letters or Stable -5-+5 letters at the annual time points
Proportion of patients that recuperate 20/20 vision (driving vision) in all patients and stratified by baseline VA (groups 1-3) | Up to 2 years
  In all patients and stratified by baseline VA (groups 1-3)
Proportion of patients that recuperate 20/40 vision (driving vision) in all patients and stratified by baseline VA (groups 1-3) | Up to 2 years
  In all patients and stratified by baseline VA (groups 1-3)
Proportion of patients with no need of Vision Aid support | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Lund, Sweden